CLINICAL TRIAL: NCT00385697
Title: A Phase 2/3, Randomized, Double-Blind, Multicenter, Multinational, 4-Arm, Controlled, Dose-Ranging Study to Evaluate Efficacy and Safety of MGA031, a Humanized, FcR Non-Binding, Anti-CD3 Monoclonal Antibody, in Children and Adults With Recent-Onset Type 1 Diabetes Mellitus
Brief Title: The Protégé Study - Clinical Trial of MGA031 in Children and Adults With Recent-Onset Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: MacroGenics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-MGA031-01
Record Dates: First submitted 2006-10-07; First posted 2006-10-11 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Randomized; Double Blind; Parallel Group; Controlled Clinical Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — teplizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Double-blind Herold Regimen (Experimental): Full dose of teplizumab IV for 14 days, repeated at Week 26
  Interventions: Biological: Teplizumab
- Double-blind 33.3% Herold Regimen (Experimental): One third full dose of teplizumab IV for 14 days, repeated at Week 26
  Interventions: Biological: Teplizumab
- Double-blind Curtailed Herold Regimen (Experimental): Full dose of teplizumab IV for 6 days followed by placebo for 8 days, repeated at Week 26
  Interventions: Biological: Teplizumab
- Double-blind Placebo (Placebo Comparator): Placebo IV dosing daily for 14 days repeated at Week 26
  Interventions: Drug: Placebo
- Open-label Herold Regimen (Experimental): Full dose of teplizumab IV for 14 days, repeated at Week 26
  Interventions: Biological: Teplizumab

INTERVENTIONS:
Biological: Teplizumab — Daily IV dosing for 14 days, repeated at Week 26
  Other Names: MGA031
  Arms: Double-blind 33.3% Herold Regimen; Double-blind Curtailed Herold Regimen; Double-blind Herold Regimen; Open-label Herold Regimen
Drug: Placebo — Daily IV dosing for 14 days, repeated at Week 26
  Arms: Double-blind Placebo

SUMMARY:
The primary purpose of this protocol is to assess the efficacy, tolerability, and safety of MGA031 when administered according to 3 different MGA031 dosing regimens in children and adults with recent-onset (diagnosis within past 12 weeks) type 1 diabetes mellitus. All regimens will be administered as an addition to insulin and other standard of care treatments. Efficacy will be defined primarily by the capacity of MGA031 to markedly reduce typical insulin requirements while maintaining relatively normal blood sugar levels.

Other studies involving the study drug use the name hOKT3γ1 (Ala-Ala). MGA031, a humanized monoclonal antibody, is the name used for hOKT3γ1 (Ala-Ala) that is produced by MacroGenics, Inc. The United States Adopted Name (USAN) for MGA031 is teplizumab.

DETAILED DESCRIPTION:
The Protégé Study - A Multinational Clinical Trial of MGA031 for Preserving the Capability to Produce Insulin, Reducing Insulin Usage and Improving Blood Sugar Levels in Children and Adults With Recent-Onset Type 1 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Enrollment (Segment #1) or randomization (Segment #2) on Study Day 0 within 12 weeks of first visit to any physician for symptoms or signs of diabetes. Study Day 0 is the first day of study drug dosing.
2. Diagnosis of type 1 diabetes mellitus, according to the American Diabetes Association (ADA) criteria
3. Requirement for injected insulin therapy
4. Have a detectable fasting or stimulated C-peptide level (above the lower limit of detection of the assay)
5. One positive result on testing for any of the following antibodies:

   1. islet-cell autoantibodies (ICA512/IA-2),
   2. glutamic acid decarboxylase autoantibodies, or
   3. insulin autoantibodies (if present during first 2 weeks, but not beyond 2 weeks, of insulin treatment)
6. Male or female
7. Subject must be in one of the following age groups:

   * Age 18-35 years
   * Age 12-17 years pending approval by Data Monitoring Committee
   * Age 8-11 years pending approval by Data Monitoring Committee
8. Body weight ≥ 36 kg

Exclusion Criteria:

Subjects must have none of the following:

1. Prior administration of a monoclonal antibody -- within the 1 year before enrollment or randomization at Study Day 0 -- that could potentially prevent or confound a therapeutic response to MGA031
2. Participation in any type of therapeutic drug or vaccine clinical trial within the 12 weeks before enrollment or randomization
3. Any medical condition that, in the opinion of the investigator, would interfere with safe completion of the trial
4. Pregnant or lactating females
5. Prior murine OKT®3 treatment at any time before enrollment or randomization
6. Current or planned therapy with exenatide or any other agents that stimulate pancreatic beta cell regeneration or insulin secretion
7. Current or planned therapy with inhaled insulin
8. Uncompensated heart failure, fluid overload, myocardial infarction or evidence of ischemic heart disease, or other serious cardiac disease within the 12 weeks before enrollment or randomization
9. History of epilepsy, cancer, cystic fibrosis, sickle cell anemia, neuropathy, peripheral vascular disease or cerebrovascular disease
10. Newly diagnosed hypothyroidism (not currently being treated but which, in the opinion of the investigator, should be treated) or active Graves' disease
11. Eczema, asthma or severe atopic disease requiring treatment within the 12 weeks before enrollment or randomization
12. Evidence of active infection, such as fever ≥ 38.0 degrees Celsius (100.5 degrees Fahrenheit)
13. Known or suspected infection with human immunodeficiency virus (HIV)
14. Evidence of active hepatitis B (HBV) or hepatitis C virus (HCV)
15. Evidence of active or latent tuberculosis
16. Vaccination with a live virus within the 8 weeks before enrollment or randomization or planned live virus vaccination continuing through week 52 of the study. Vaccination with an antigen or killed organism must not be given within 8 weeks before or planned within 8 weeks after each dosing cycle.
17. Any infectious mononucleosis-like illness within the 6 months before enrollment or randomization
18. Serologic and clinical evidence of acute infection with Epstein-Barr virus (EBV)
19. Serologic evidence of acute infection with cytomegalovirus (CMV)

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 554 (Actual)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (115):
- United States (39):
  - UAB School of Medicine, Birmingham, Alabama
  - NEA Clinic, Jonesboro, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Diabetes Medical Center of California, Northridge, California
  - UCSF Medical Center, San Francisco, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Christiana Care Research Institute, Newark, Delaware
  - Richard Hays, MD, Wellington, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Humphrey Diabetes Center, Boise, Idaho
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Mid-America Diabetes Associates, PA, Wichita, Kansas
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - St. Agnes Hospital, Baltimore, Maryland
  - Maryland Diabetes & Endocrine Associates, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Alzohaili Medical Consultants, Dearborn, Michigan
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Creighton Diabetes Center, Omaha, Nebraska
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - University of Medicine & Dentistry of NJ, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Joslin Diabetes Center, Syracuse, New York
  - Cleveland Clinic, Cleveland, Ohio
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Sumter Medical Specialists, Sumter, South Carolina
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - Methodist Healthcare, Memphis, Tennessee
  - Research Institute of Dallas, Dallas, Texas
  - Spectra Research Center, McAllen, Texas
  - Diabetes and Glandular Disease Research, San Antonio, Texas
  - Endocrine Research Specialists, Ogden, Utah
  - Pacific Northwest Research Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - University Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Capital District Health Authority, Halifax, Nova Scotia
  - Oxford AIM Clinic, London, Ontario
  - Children's Hospital of Western, London, Ontario
- Czechia (6):
  - FN Brno- Detska nemocnice, Brno
  - FN Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - FN Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
  - Masarykova nemocnice v Usti nad Labem, Ústí nad Labem
- Estonia (2):
  - Tartu University Hospital, Puusepa, Tartu
  - East Tallinn Central Hospital, Tallinn
- Germany (5):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Medizinische Universitätsklinik Ulm, Ulm, Baden-Wurttemberg
  - Herz-und Diabetszentrum Nordrhein-Westfalen, Bad Oeynhausen, North Rhine-Westphalia
  - Charité-Hochschulmedizin Berlin, Berlin
  - Universitatsklinik Giessen, Giessen
- India (15):
  - Nizam's Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Gujarat Endocrine Centre, Ahmedabad, Gujarat
  - DHL Research Centre, Ahmedabad, Gujarat
  - Bharti Research Institute of Diabetes & Endocrinology, Karnāl, Haryana
  - Bangalore Diabetes Centre, Bangalore, Karnataka
  - Diabetes Thyroid Hormone Research Institute PVT LTD, Indore, Madhya Pradesh
  - Diabetes Action Centre, Mumbai, Maharashtra
  - Gandhi Endocrinology and Diabetes Centre, Nagpur, Maharashtra
  - Endocrine Clinic, Nashik, Maharashtra
  - Grant Medical Foundation, Pune, Maharashtra
  - Fortis Escorts Hospital, Jaipur, Rajasthan
  - B.P.Poddar Hospital and Medical Research Ltd, Kolkata, West Bengal
  - Medwin Hospitals, Hyderabad
  - Pushpawati Singhania Research Institute, New Delhi
- Israel (6):
  - Soroka Medical Centre, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Centre, Haifa
  - Wolfson Medical Centre, Holon
  - National Centre for Childhood and Diabetes, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- P. Stradins Clinical University Hospital, Riga, Latvia
- Mexico (4):
  - Hospital CIMA Santa Engracia, San Pedro Garza García, Nuevo León
  - Hospital Mexico-Americano, Guadalajara
  - Hospital General de Mexico, Mexico City
  - Hospital Central, San Luis Potosí City
- Diabeter Center for Pediatric and Adolescent Diabetes Care and Research, Rotterdam, Netherlands
- Poland (7):
  - Samodzielny Publiczny Szpital Kliniczny Akademi Medycznej w Bialymstoku, Bialystok
  - Oddzial Diabetologiczny Klinika Pediatrii, Gdansk
  - Wojewodzki Specjalistyczny Szpital Dzieciecy, Kielce
  - Uniwersytecki Szpital Kliniczny, Lodz
  - I. Szpital Miejski im. Dr. E. Sonnenberga w Lodzi, Lodz
  - Powiatowy Zespot Szpitali w Olesnicy, Oddzial Chorob Wewnetrznych, Oleśnica
  - Klinika Endokrynologii i Diabetologii Wieku Rozwojowego, Wroclaw
- Romania (6):
  - S.C. Minimed S.R.L., Bacau
  - Institutul de Diabet, Bucharest
  - Centrul Medical "Sanatatea ta", Bucharest
  - Spitulul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta, Iași
  - Spitalul Judetean Satu Mare, Satu Mare
- Spain (5):
  - Hospital Universitari Dr. Josep Trueta de Girona, Girona, Gerona
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic I Provincial, Barcelona
  - Fundacion Jimenez Diaz, Madrid
- Sweden (3):
  - Universitetssjukhuset i Linkoping, Linköping
  - Universitetssjukhuset i Lund, Lund
  - Sodersjukhuset AB, Stockholm
- Ukraine (7):
  - Donetsk Regional Children Clinical Hospital, Donetsk
  - V. Danilevsky Institute of Endocrine Pathology Problems, Kharkiv
  - Kharkiv Regional Clinical Children's Hospital, Kharkiv
  - Ukrainian Scientific and Practical Center of Endocrine Surgery, Kyiv
  - Ukranian Children Specialised Clinical Hospital, Kyiv
  - Regional Clinical Endocrinological Dispensary, Vinnitsa
  - Zaporizhzhya Regional Pediatric Hospital, Zaporizhzhya
- United Kingdom (2):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Royal Devon and Exeter Hospital, Exeter, Devon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417
- [Derived] Sherry N, Hagopian W, Ludvigsson J, Jain SM, Wahlen J, Ferry RJ Jr, Bode B, Aronoff S, Holland C, Carlin D, King KL, Wilder RL, Pillemer S, Bonvini E, Johnson S, Stein KE, Koenig S, Herold KC, Daifotis AG; Protege Trial Investigators. Teplizumab for treatment of type 1 diabetes (Protege study): 1-year results from a randomised, placebo-controlled trial. Lancet. 2011 Aug 6;378(9790):487-97. doi: 10.1016/S0140-6736(11)60931-8. Epub 2011 Jun 28. PMID 21719095

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Herold Regimen; Double-blind Herold Regimen: Full dose of teplizumab IV for 14 days, repeated at Week 26 Teplizumab: Daily IV dosing for 14 days, repeated at Week 26
- Double-blind Placebo: Placebo IV dosing daily for 14 days repeated at Week
  Placebo: Daily IV dosing for 14 days, repeated at Week 26
Period: Open-label Segment 1
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Started | 38 | 0 | 0 | 0 | 0
Completed | 35 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Period: Double-blind Segment 2
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Started | 0 | 209 (2 patients were randomized but not dosed, so are not included in baseline demographics or region of enrollment.) | 102 | 106 | 99 (1 patient was randomized and not dosed, so not included in baseline demographics or region of enrollment..)
Full Analysis Set (FAS) Population (Randomized subjects that received any amount of study treatment, analyzed according to randomization.) | 0 | 207 | 102 | 106 | 98
Safety Population (Randomized subjects that received any amount of study treatment, analyzed according to actual treatment received.) | 0 | 207 | 102 | 106 | 98
Completed | 0 | 183 | 90 | 97 | 92
Not Completed | 0 | 26 | 12 | 9 | 7
Not completed — Adverse Event | 0 | 3 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 11 | 5 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 10 | 6 | 7 | 2
Not completed — Other | 0 | 2 | 0 | 0 | 0
Period: Long-term Follow up Segment 3
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Started | 35 | 183 | 90 | 97 | 92
Completed | 35 | 183 | 90 | 97 | 92
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for age, six, race and ethnicity are from the FAS, which includes only those participants enrolled and receiving study treatment (n=551). There were 3 participants enrolled who were never dosed so they are excluded from the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo | Total
Number analyzed (Participants) | 38 | 209 | 102 | 106 | 99 | 554
Age, Continuous [Median (Full Range); unit: years] — Population: Baseline characteristics for age, six, race and ethnicity are from the FAS, which includes only those participants enrolled and receiving study treatment (n=551). There were 3 participants enrolled who were never dosed so they are excluded from the FAS.
  years
    number analyzed (Participants) | 38 | 207 | 102 | 106 | 98 | 551
    (all) | 13.5 [10.0 to 34.0] | 17 [8 to 35] | 17 [8 to 34] | 16 [8 to 33] | 17 [8 to 34] | 17 [8 to 35]
Age, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics for age, six, race and ethnicity are from the FAS, which includes only those participants enrolled and receiving study treatment (n=551). There were 3 participants enrolled who were never dosed so they are excluded from the FAS.
  Participants
    number analyzed (Participants) | 38 | 207 | 102 | 106 | 98 | 551
    age 8-11 years | 11 | 31 | 15 | 16 | 15 | 88
    age 12-17 years | 16 | 81 | 42 | 44 | 38 | 221
    age 18-35 years | 11 | 95 | 45 | 46 | 45 | 242
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics for age, six, race and ethnicity are from the FAS, which includes only those participants enrolled and receiving study treatment (n=551). There were 3 participants enrolled who were never dosed so they are excluded from the FAS.
  Participants
    number analyzed (Participants) | 38 | 207 | 102 | 106 | 98 | 551
    Female | 8 | 77 | 40 | 34 | 37 | 196
    Male | 30 | 130 | 62 | 72 | 61 | 355
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics for age, six, race and ethnicity are from the FAS, which includes only those participants enrolled and receiving study treatment (n=551). There were 3 participants enrolled who were never dosed so they are excluded from the FAS.
  Participants
    number analyzed (Participants) | 38 | 207 | 102 | 106 | 98 | 551
    Hispanic or Latino | 2 | 14 | 7 | 12 | 5 | 40
    Not Hispanic or Latino | 36 | 193 | 95 | 94 | 93 | 511
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics for age, six, race and ethnicity are from the FAS, which includes only those participants enrolled and receiving study treatment (n=551). There were 3 participants enrolled who were never dosed so they are excluded from the FAS.
  Participants
    number analyzed (Participants) | 38 | 207 | 102 | 106 | 98 | 551
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 5 | 59 | 28 | 29 | 27 | 148
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 1 | 1 | 2
    White | 33 | 145 | 74 | 75 | 69 | 396
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 3 | 0 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants] — The data on region of enrollment is based on the total number of patients started, n=554.
  participants
    Romania | 4 | 7 | 5 | 4 | 4 | 24
    United States | 20 | 64 | 32 | 31 | 31 | 178
    Czechia | 8 | 12 | 7 | 5 | 6 | 38
    Ukraine | 0 | 18 | 10 | 9 | 10 | 47
    Spain | 0 | 6 | 3 | 3 | 3 | 15
    India | 5 | 59 | 28 | 29 | 28 | 149
    Canada | 1 | 6 | 1 | 4 | 1 | 13
    Sweden | 0 | 0 | 0 | 1 | 0 | 1
    Latvia | 0 | 3 | 1 | 2 | 1 | 7
    Poland | 0 | 10 | 5 | 6 | 4 | 25
    Mexico | 0 | 9 | 4 | 5 | 4 | 22
    Israel | 0 | 11 | 6 | 6 | 6 | 29
    Germany | 0 | 2 | 0 | 0 | 0 | 2
    Estonia | 0 | 2 | 0 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects in Segment 2 With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and Hemoglobin A1c (HbA1c) Level of Less Than 6.5%.
Description: This is a composite endpoint is based on the proportion of subjects who have both a total daily insulin dose <0.5 U/Kg/day and an HbAlc level 6.5% at 52 weeks after randomization.
Time Frame: 52 weeks after randomization
Population: Efficacy analysis was performed on the FAS population from the double-blind Segment 2. No efficacy analysis was performed on the Open-label Segment 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 0 | 207 | 102 | 106 | 98
Participants |  | 41 | 14 | 22 | 20
Statistical Analysis 1: Comparison: Double-blind Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.904, Mantel Haenszel; Odds Ratio (OR) = 0.963, 95% CI 2-sided [0.521 to 1.779]
Statistical Analysis 2: Comparison: Double-blind 33.3% Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.222, Mantel Haenszel; Odds Ratio (OR) = 0.629, 95% CI 2-sided [0.297 to 1.330]
Statistical Analysis 3: Comparison: Double-blind Curtailed Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.885, Mantel Haenszel; Odds Ratio (OR) = 1.054, 95% CI 2-sided [0.521 to 2.129]

2. Primary Outcome: Number of Subjects in Segment 1 With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and Hemoglobin A1c (HbA1c) Level of Less Than 6.5%.
Description: This is a composite endpoint based on the proportion of subjects who have both a total daily insulin dose <0.5 U/Kg/day and an HbAlc level 6.5%
Time Frame: 52 weeks after first dose
Population: Open-label Segment 1. Participants with missing data were considered non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen
Number analyzed (Participants) | 38
Participants | 11

3. Primary Outcome: Mean HbA1c Change From Baseline in Segment 2
Description: Comparison among study treatments of average change from baseline HbA1C. This endpoint will be assessed in a hierarchical manner only if the composite primary endpoint shows a statistically significant difference between arms
Time Frame: 52 weeks after randomization
Population: Per the Analysis Plan, the change from baseline (CFB) analysis was performed on the FAS population in Double-blind Segment 2 only. The number of participants analyzed includes all participants with baseline HbA1c data at baseline and at 52 weeks after randomization. Eight participants did not have 52 week data. The analysis was not conducted for the open-label Herold Regimen because there was no placebo control.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 0 | 201 | 100 | 106 | 98
percentage of HbA1c |  | -0.42 (2.285) | -0.34 (2.196) | -0.36 (2.132) | -0.43 (2.668)
Statistical Analysis 1: Comparison: Double-blind Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.814, ANCOVA; Mean Difference (Final Values) = 0.061, 95% CI 2-sided [-0.450 to 0.572]
Statistical Analysis 2: Comparison: Double-blind 33.3% Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.593, ANCOVA; Mean Difference (Final Values) = 0.161, 95% CI 2-sided [-0.433 to 0.755]
Statistical Analysis 3: Comparison: Double-blind Curtailed Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.886, ANCOVA; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.594 to 0.513]

4. Primary Outcome: Mean HbA1c Change From Baseline in Segment 1
Description: The average change in HbA1c levels after dosing.
Time Frame: 52 weeks after first dose
Population: Open-label Segment 1.
Measure: Mean (Standard Deviation); unit: percent HbA1c
Arm/Group | Open-label Herold Regimen
Number analyzed (Participants) | 38
percent HbA1c | 0.25 (2.053)

5. Secondary Outcome: Change From Baseline in C-peptide Area Under the Curve (AUC) in Segment 2
Description: Comparison among study treatments on the AUC of C-peptide secretory responses following a mixed meal eaten by the subject
Time Frame: 104 weeks after randomization
Population: Per the Analysis Plan, the change from baseline (CFB) analysis was performed on the FAS population in Double-blind Segment 2 only. The number of participants analyzed includes all participants with baseline C-peptide data at baseline and at 52 weeks after randomization. Eight participants did not have 52 week data. The analysis was not conducted for the open-label Herold Regimen because there was no placebo control.
Measure: Mean (Standard Deviation); unit: min*nmol/L
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 0 | 201 | 100 | 102 | 96
min*nmol/L |  | -0.18 (0.355) | -0.27 (0.318) | -0.20 (0.354) | -0.22 (0.428)
Statistical Analysis 1: Comparison: Double-blind Herold Regimen; Test type: Superiority; p = 0.049, ANCOVA; Mean Difference (Final Values) = 0.047, 95% CI 2-sided [0.000 to 0.093]
Statistical Analysis 2: Comparison: Double-blind 33.3% Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.937, ANCOVA; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.061 to 0.056]
Statistical Analysis 3: Comparison: Double-blind Curtailed Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.382, ANCOVA; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.032 to 0.084]

6. Secondary Outcome: Change From Baseline in C-peptide AUC in Segment 1
Description: AUC of C-peptide secretory responses following a mixed meal eaten by the subject
Time Frame: 104 weeks after first dose
Population: Open-label Segment 1.
Measure: Mean (Standard Deviation); unit: min*nmol/L
Arm/Group | Open-label Herold Regimen
Number analyzed (Participants) | 38
min*nmol/L | -0.45 (0.451)

7. Secondary Outcome: Number of Subjects in Segment 2 With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and HbA1c Level of Less Than 6.5%
Description: Comparison among study treatments of a composite endpoint based on the proportion of subjects who have both a total daily insulin dose <0.5 U/Kg/day and an HbAlc level 6.5%.
Time Frame: 104 weeks after randomization
Population: Analysis performed on the FAS population in Double-blind Segment 2. Missing values were counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 0 | 207 | 102 | 106 | 98
Participants |  | 17 | 6 | 10 | 9
Statistical Analysis 1: Comparison: Double-blind Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.775, Mantel Haenszel; Odds Ratio (OR) = 0.881, 95% CI 2-sided [0.372 to 2.089]
Statistical Analysis 2: Comparison: Double-blind 33.3% Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.402, Mantel Haenszel; Odds Ratio (OR) = 0.628, 95% CI 2-sided [0.212 to 1.861]
Statistical Analysis 3: Comparison: Double-blind Curtailed Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.859, Mantel Haenszel; Odds Ratio (OR) = 1.093, 95% CI 2-sided [0.410 to 2.912]

8. Secondary Outcome: Number of Subjects in Segment 1 With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and HbA1c Level of Less Than 6.5%
Description: as for outcome 7
Time Frame: 104 weeks after first dose
Population: Open-label Segment 1. Participants with missing values were counted as non-responders
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen
Number analyzed (Participants) | 38
Participants | 5

9. Secondary Outcome: Number of Subjects in Segment 2 With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and HbA1c Level of Less Than 7.0%.
Description: Comparison among study treatments of a composite endpoint based on the proportion of subjects who have both a total daily insulin dose <0.5 U/Kg/day and an HbAlc level 7.0%.
Time Frame: at 52 weeks after randomization
Population: Analysis performed on the FAS population in Double-blind Segment 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 0 | 207 | 102 | 106 | 98
Participants |  | 60 | 21 | 28 | 24
Statistical Analysis 1: Comparison: Double-blind Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.404, Mantel Haenszel; Odds Ratio (OR) = 1.265, 95% CI 2-sided [0.727 to 2.200]
Statistical Analysis 2: Comparison: Double-blind 33.3% Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.528, Mantel Haenszel; Odds Ratio (OR) = 0.805, 95% CI 2-sided [0.412 to 1.576]
Statistical Analysis 3: Comparison: Double-blind Curtailed Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.706, Mantel Haenszel; Odds Ratio (OR) = 1.133, 95% CI 2-sided [0.594 to 2.164]

10. Secondary Outcome: Number of Subjects in Segment 1 With Both a Total Daily Insulin Dose of Less Than 0.5 U/kg/Day and HbA1c Level of Less Than 7.0%.
Description: Composite endpoint based on the proportion of subjects who have both a total daily insulin dose <0.5 U/Kg/day and an HbAlc level 7.0%.
Time Frame: 52 weeks after first dose
Population: Open-label Segment 1. Missing values counted as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Herold Regimen
Number analyzed (Participants) | 38
Participants | 14

11. Secondary Outcome: Mean HbA1c Change From Baseline in Segment 2
Description: Comparison among study treatments of the average change from baseline in HbA1c.
Time Frame: at 104 weeks after randomization
Population: Per the Analysis Plan, the change from baseline (CFB) analysis was performed on data available for the FAS population in Double-blind Segment 2 only. The analysis was not conducted for the open-label Herold Regimen because there was no placebo control.
Measure: Mean (Standard Deviation); unit: percent of HbA1c
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
Number analyzed (Participants) | 0 | 201 | 100 | 106 | 98
percent of HbA1c |  | 0.14 (2.411) | 0.08 (2.261) | 0.04 (2.208) | 0.16 (2.510)
Statistical Analysis 1: Comparison: Double-blind Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.872, ANCOVA; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [-0.455 to 0.536]
Statistical Analysis 2: Comparison: Double-blind 33.3% Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.979, ANCOVA; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.581 to 0.556]
Statistical Analysis 3: Comparison: Double-blind Curtailed Herold Regimen vs Double-blind Placebo; Test type: Superiority; p = 0.400, ANCOVA; Mean Difference (Final Values) = -0.225, 95% CI 2-sided [-0.750 to 0.301]

12. Secondary Outcome: Mean HbA1c Change From Baseline in Segment 1
Description: Comparison among study treatments of the average change from baseline in HbA1c.
Time Frame: 104 weeks after first dose
Population: Analysis performed on the FAS population in Double-blind Segment 2
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Open-label Herold Regimen
Number analyzed (Participants) | 38
percentage of HbA1c | 0.73 (2.091)

ADVERSE EVENTS:
Time Frame: Adverse events (AE), serious adverse events (SAE), and adverse events of special interest (AESI) were collected through Week 52. Only SAE and AESI were collected after Week 53 through Week 104.
Arm/Group | Open-label Herold Regimen | Double-blind Herold Regimen | Double-blind 33.3% Herold Regimen | Double-blind Curtailed Herold Regimen | Double-blind Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 1/207 | 1/102 | 0/106 | 0/98
Serious Adverse Events (participants affected / at risk) | 6/38 | 23/207 | 14/102 | 12/106 | 12/98
Other Adverse Events (participants affected / at risk) | 38/38 | 207/207 | 101/102 | 105/106 | 98/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Herold Regimen (N=38) | Double-blind Herold Regimen (N=207) | Double-blind 33.3% Herold Regimen (N=102) | Double-blind Curtailed Herold Regimen (N=106) | Double-blind Placebo (N=98)
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 — inflammation of throat and tonsils
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 6 | 3 | 2 | 0 — Too many ketones in the bloodstream
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 1 — Too much sugar in the bloodstream
Ketonuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 — Ketones in the urine
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 — Not enough infection fighting blood cells
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 — heart attack
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 1 | 0 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0 — Fever
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 2
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 — abnormal gallbladder function
Biloma (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 — a collection of bile outside the gallbladder
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 — inflammation of the gallbladder
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 — enlarged liver and spleen
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 — Stomach flu
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 1 | 0 — Stomach flu
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Renal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 — severe infection in the bloodstream
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 — skin infection
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 — nail inflammation
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Ketosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Intercapillary glomerulosclerosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 — degenerative disease in the kidney due to diabetes
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 — abnormal albumin in the urine
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 — Epididymitis is swelling or pain in the back of the testicle in the coiled tube (epididymis) that stores and carries sperm.
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 — blood clot in the subclavian vein
Keytonuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 — Too many ketones in the urine
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Herold Regimen (N=38) | Double-blind Herold Regimen (N=207) | Double-blind 33.3% Herold Regimen (N=102) | Double-blind Curtailed Herold Regimen (N=106) | Double-blind Placebo (N=98)
Lymphopenia (Blood and lymphatic system disorders) | 36 | 152 | 67 | 81 | 17 — low lymphocyte count
Leukopenia (Blood and lymphatic system disorders) | 25 | 101 | 49 | 50 | 22 — low white blood cell count
Neutropenia (Blood and lymphatic system disorders) | 15 | 71 | 33 | 22 | 18 — low neutrophil count
Anaemia (Blood and lymphatic system disorders) | 4 | 29 | 13 | 8 | 10 — low red blood cell count
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 22 | 8 | 16 | 10 — low platelet count
Nausea (Gastrointestinal disorders) | 9 | 41 | 15 | 21 | 12
Vomiting (Gastrointestinal disorders) | 8 | 30 | 6 | 14 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 13 | 6 | 6 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 10 | 4 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 10 | 2 | 2 | 5
Pyrexia (General disorders) | 9 | 42 | 18 | 28 | 21 — Fever
Fatigue (General disorders) | 3 | 22 | 9 | 15 | 6
Application site rash (General disorders) | 2 | 2 | 0 | 3 | 0
Asthenia (General disorders) | 2 | 7 | 4 | 4 | 3
Catheter site pain (General disorders) | 2 | 1 | 1 | 2 | 3
Chills (General disorders) | 2 | 20 | 5 | 13 | 2
Hyperbilirubinemia (Hepatobiliary disorders) | 5 | 25 | 11 | 8 | 9 — elevated blood bilirubin
Cytokine release syndrome (Immune system disorders) | 3 | 12 | 3 | 9 | 0
Seasonal allergy (Immune system disorders) | 2 | 5 | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 30 | 20 | 22 | 15
Nasopharyngitis (Infections and infestations) | 3 | 28 | 11 | 15 | 13
Pharyngitis (Infections and infestations) | 2 | 11 | 8 | 4 | 3 — throat inflammation
Sinusitis (Infections and infestations) | 4 | 8 | 7 | 6 | 7
Influenza (Infections and infestations) | 1 | 11 | 4 | 5 | 8
Rhinitis (Infections and infestations) | 1 | 9 | 5 | 4 | 5 — Runny nose
Otitis media (Infections and infestations) | 2 | 3 | 2 | 1 | 3 — ear infection
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 13 | 92 | 60 | 41 | 38
White blood cell count decreased (Investigations) | 15 | 86 | 32 | 41 | 18
Aspartate aminotransferase increased (Investigations) | 17 | 73 | 28 | 37 | 33
Alanine aminotransferase increased (Investigations) | 16 | 71 | 26 | 31 | 17
Haemoglobin decreased (Investigations) | 14 | 66 | 29 | 34 | 32
Lymphocyte count decreased (Investigations) | 6 | 49 | 14 | 25 | 9
Blood sodium decreased (Investigations) | 5 | 43 | 20 | 19 | 17
Neutrophil count decreased (Investigations) | 11 | 40 | 18 | 24 | 15
Blood alkaline phosphatase increased (Investigations) | 7 | 31 | 16 | 14 | 22
Platelet count decreased (Investigations) | 4 | 34 | 12 | 15 | 9
Blood bilirubin increased (Investigations) | 4 | 17 | 9 | 7 | 5
Bilirubin conjugated increased (Investigations) | 1 | 17 | 6 | 5 | 2
Gamma-glutamyltransferase increased (Investigations) | 4 | 10 | 7 | 7 | 10
Blood calcium decreased (Investigations) | 2 | 25 | 14 | 14 | 9
Blood albumin decreased (Investigations) | 3 | 23 | 6 | 9 | 5
Blood potassium decreased (Investigations) | 3 | 11 | 8 | 9 | 6
Blood phosphorus decreased (Investigations) | 1 | 11 | 6 | 10 | 7
Blood potassium increased (Investigations) | 2 | 8 | 9 | 5 | 5
Blood creatinine increased (Investigations) | 3 | 6 | 7 | 9 | 3
Blood phosphorus increased (Investigations) | 2 | 9 | 7 | 4 | 5
Eosinophil count increased (Investigations) | 4 | 6 | 2 | 4 | 2
Haematocrit decreased (Investigations) | 4 | 9 | 4 | 10 | 8
Blood urea increased (Investigations) | 3 | 4 | 4 | 5 | 4
Epstein-Barr virus antibody positive (Investigations) | 3 | 6 | 4 | 1 | 5
Blood calcium increased (Investigations) | 3 | 6 | 5 | 3 | 5
Blood glucose increased (Investigations) | 2 | 0 | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 10 | 4 | 10 | 9
Haemoglobin increased (Investigations) | 3 | 1 | 0 | 0 | 0
Monocyte count increased (Investigations) | 3 | 2 | 0 | 0 | 0
Haematocrit increased (Investigations) | 2 | 1 | 0 | 0 | 1
Mean cell haemoglobin decreased (Investigations) | 2 | 0 | 1 | 2 | 2
Mean cell volume decreased (Investigations) | 2 | 1 | 0 | 3 | 0
Neutrophil count increased (Investigations) | 2 | 2 | 0 | 2 | 2
Red blood cell count increased (Investigations) | 2 | 0 | 1 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 64 | 35 | 38 | 34
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 57 | 18 | 30 | 25
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 22 | 14 | 13 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 20 | 10 | 13 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 14 | 8 | 10 | 10
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 16 | 6 | 5 | 6
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 9 | 6 | 4 | 9 — too much sodium in the bloodstream
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 5 | 1
Headache (Nervous system disorders) | 10 | 53 | 25 | 26 | 17
Dizziness (Nervous system disorders) | 1 | 10 | 3 | 5 | 6
Proteinuria (Renal and urinary disorders) | 8 | 24 | 17 | 12 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 17 | 7 | 8 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 18 | 5 | 3 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 5 | 5 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 2 | 3 — runny nose
Rash (Skin and subcutaneous tissue disorders) | 17 | 65 | 44 | 37 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 4 | 0 | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 2 | 0 — increased sweating
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 32 | 10 | 12 | 4 — Itching
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 11 | 3 | 5 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 4 | 5
Goitre (Endocrine disorders) | 2 | 3 | 0 | 2 | 3 — irregular growth of the thyroid gland
Influenza like illness (General disorders) | 0 | 5 | 3 | 1 | 5
Blood chloride increased (Investigations) | 1 | 7 | 4 | 7 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 10 | 7 | 8 | 4 — too little phosphate in the blood
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 6 | 3 | 2 — joint pain
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 6 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 3 | 2 | 3 | 3 — Stomach flu
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less